CLINICAL TRIAL: NCT07064018
Title: Phase Ib/IIa Trial of Single Protein Encapsulated Doxorubicin, SPEDOX-6 in Advanced Malignancies
Brief Title: Trial of Single Protein Encapsulated Doxorubicin, SPEDOX-6 in Advanced Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Sunstate Biosciences LLC (Industry)
Responsible Party: Principal Investigator, Warren Chow, Professor - Division of Hematology-Oncology, Department of Medicine, UCI School of Medicine, University of California, Irvine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 6228; UCI 24-08 (Other: UCI CFCCC)
Record Dates: First submitted 2025-05-27; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Soft-tissue Sarcoma; Triple Negative Breast Cancer; Non-small Cell Lung Cancer; Cervical Cancer; Ovarian Cancer; KRAS Mutation-Related Tumors
MeSH Terms: conditions — Sarcoma; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms; Ovarian Neoplasms | interventions — pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Phase 1b Dose Level 1 - Spedox-6 (Experimental): Spedox-6, 20 mg/m2, Chemotherapy single agent systemic, received on day 1 of each 21 day cycle, for a total of 6 cycles.
  Interventions: Drug: Spedox-6
- Phase 1b Dose Level 2 - Spedox-6 + Filgrastim/Pegfilgrastim (Experimental): Spedox-6, 40 mg/m2, Chemotherapy single agent systemic, received on day 1 of each 21 day cycle, for a total of 6 cycles.
  Filgrastim or Pegfilgrastin, injected subcutaneously or intravenously, received according to Institutional standard.
  Interventions: Drug: Spedox-6; Drug: Pegfilgrastim; Drug: Filgrastim
- Phase 1b Dose Level 3 - Spedox-6 + Filgrastim/Pegfilgrastim (Experimental): Spedox-6, 80 mg/m2, Chemotherapy single agent systemic, received on day 1 of each 21 day cycle, for a total of 6 cycles.
  Filgrastim or Pegfilgrastin, injected subcutaneously or intravenously, received according to Institutional standard.
  Interventions: Drug: Spedox-6; Drug: Pegfilgrastim; Drug: Filgrastim
- Phase 1b Dose Level 4 - Spedox-6 + Filgrastim/Pegfilgrastim (Experimental): Spedox-6, 120 mg/m2, Chemotherapy single agent systemic, received on day 1 of each 21 day cycle, for a total of 6 cycles.
  Filgrastim or Pegfilgrastin, injected subcutaneously or intravenously, received according to Institutional standard.
  Interventions: Drug: Spedox-6; Drug: Pegfilgrastim; Drug: Filgrastim
- Phase 1b Dose Level 5 - Spedox-6 + Filgrastim/Pegfilgrastim (Experimental): Spedox-6, 160 mg/m2, Chemotherapy single agent systemic, received on day 1 of each 21 day cycle, for a total of 6 cycles.
  Filgrastim or Pegfilgrastin, injected subcutaneously or intravenously, received according to Institutional standard.
  Interventions: Drug: Spedox-6; Drug: Pegfilgrastim; Drug: Filgrastim
- Phase 1b Dose Level 6 - Spedox-6 + Filgrastim/Pegfilgrastim (Experimental): Spedox-6, 200 mg/m2, Chemotherapy single agent systemic, received on day 1 of each 21 day cycle, for a total of 6 cycles.
  Filgrastim or Pegfilgrastin, injected subcutaneously or intravenously, received according to Institutional standard.
  Interventions: Drug: Spedox-6; Drug: Pegfilgrastim; Drug: Filgrastim
- Phase 1b Dose Level 7 - Spedox-6 + Filgrastim/Pegfilgrastim (Experimental): Spedox-6, 250 mg/m2, Chemotherapy single agent systemic, received on day 1 of each 21 day cycle, for a total of 6 cycles.
  Filgrastim or Pegfilgrastin, injected subcutaneously or intravenously, received according to Institutional standard.
  Interventions: Drug: Spedox-6; Drug: Pegfilgrastim; Drug: Filgrastim
- Phase 1b Dose Level 8 - Spedox-6 + Filgrastim/Pegfilgrastim (Experimental): Spedox-6, 310 mg/m2, Chemotherapy single agent systemic, received on day 1 of each 21 day cycle, for a total of 6 cycles.
  Filgrastim or Pegfilgrastin, injected subcutaneously or intravenously, received according to Institutional standard.
  Interventions: Drug: Spedox-6; Drug: Pegfilgrastim; Drug: Filgrastim

INTERVENTIONS:
Drug: Spedox-6 — Given Intravenously (IV)
Drug: Pegfilgrastim — Given Subcutaneous Injection or IV
  Arms: Phase 1b Dose Level 2 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 3 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 4 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 5 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 6 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 7 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 8 - Spedox-6 + Filgrastim/Pegfilgrastim
Drug: Filgrastim — Given Subcutaneous Injection or IV
  Arms: Phase 1b Dose Level 2 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 3 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 4 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 5 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 6 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 7 - Spedox-6 + Filgrastim/Pegfilgrastim; Phase 1b Dose Level 8 - Spedox-6 + Filgrastim/Pegfilgrastim

SUMMARY:
This is a Phase 1b/IIa dose escalation clinical trial determining the recommended phase II dose of SPEDOX-6 in subjects with advanced, therapy-refractory soft-tissue sarcoma (STS); triple-negative breast cancer (TNBC); Non-small cell lung cancer (NSCLC); cervical cancer; ovarian cancer; KRAS mutant pancreatic ductal adenocarcinoma. These are subjects who have not previously been treated with anthracyclines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years at the first screening examination/visit.
* Subjects with advanced histologically or cytologically confirmed solid tumors (see below) refractory to or relapse from at least two previous therapies.
* Tumor types expected to express lower levels of FcRn relative to normal tissue including: STS, TNBC, cervical cancer, NSCLC, ovarian cancer, and KRAS mutated pancreatic ductal adenocarcinoma without requirement for testing FcRn level.
* Disease that is considered measurable by RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Life expectancy of at least 12 weeks.
* Human Immunodeficiency Virus (HIV)-positive trial participants should be on established antiretroviral therapy (ART) for at least four weeks and have an HIV viral load less than 400 copies/mL prior to enrollment.
* Left ventricular ejection fraction > 50%.
* Adequate organ function: (Hb ≥10 g/dL, ANC ≥1,000/µL3, and platelets

  ≥100,000/µL3), serum bilirubin ≤.5x the institutional upper limit of normal (ULN) (unless known Gilbert's disease), Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤3x ULN, and creatinine clearance >50 mL/min as assessed by Cockcroft-Gault equation.
* For patients with known Gilbert's disease, serum unconjugated bilirubin must be < 4 mg/dL.
* Patient must have washed out of prior chemotherapy (at least 3 weeks from last end of therapy), radiotherapy (at least 4 weeks from last end of therapy), immunotherapy (at least 4 weeks from last end of therapy), other targeted therapies (at least 4 weeks from last end of therapy), or surgery (at least 4 weeks).
* Recovery from toxicities of prior therapy. Toxicities should have recovered to CTCAE grade ≤ 1 or baseline with exception of alopecia.
* Females of reproductive potential must have had a negative pregnancy test performed within 7 days prior to the start of treatment. Additionally, female subjects of reproductive potential should agree to use effective acceptable forms of contraception: surgical sterilization (tubal ligation); total abstinence from sexual intercourse with the opposite sex; established hormonal birth control (e.g., oral, transdermal, injection, or implant) plus a barrier method or a double barrier method (intrauterine device, spermicide, or a diaphragm plus condom) for at least 1 month prior to Cycle 1 Day 1 and agreement to use such a method during study participation and for an additional 6 months after the last dose of SPEDOX-6.
* For males of reproductive potential: vasectomy or highly effective contraception (e.g., condoms, abstinence) during the study and for an additional 6 months after the last dose of SPEDOX-6.

Exclusion Criteria:

* Patients with cancers with known driver mutations for which there are known and effective targeted therapies that have not received those therapies, but are able to. If a patient has received appropriate targeted treatment for their mutations and progressed, or those treatments are contraindicated, they will be considered potentially eligible.
* Unstable angina pectoris, angioplasty, cardiac stenting, or myocardial infarction 6 months before study entry.
* Untreated metastases to the Central Nervous System (CNS).
* Have received any prior doxorubicin or anthracycline equivalent.
* Previous radiation to the mediastinal or pericardial area.
* A known allergy to albumin.
* HIV infection with CD4+ count < 350 cells/µL or Acquired Immunodeficiency (AIDS)-defining opportunistic infection in previous 12 months.
* Pregnant (positive serum or urine pregnancy test) or lactating.
* Previous treatment with an investigational agent or the non-approved use of a drug or device withing 4 weeks of study entry.
* Uncontrolled diabetes mellitus.
* Patients who require concomitant use of strong inhibitors or inducers of CYP3A4, CYP2D6 or P-glycoprotein (P-gp).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) by RECIST v1.1 | 2 Years
  Sum of Complete Response (CR) and Partial Response (PR) by RECIST v1.1. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1): Complete Response (CR) is defined as the disappearance of all target lesions; Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions. ORR = CR + PR
Disease Control Rate (DCR) by RECIST v1.1 | 2 Years
  Disease Control Rate (DCR) defined as Sum of Stable Disease (SD) + Partial Response (PR) + Complete Response (CR) by RECIST v1.1. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1): Complete Response (CR) is defined as the disappearance of all target lesions; Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD is defined as an increase of at least 20% in the sum of the longest diameters of the target lesions, with an absolute increase of at least 5 mm, or the appearance of one or more new lesions. Stable Disease (SD) is defined as a tumor that has neither shrunk sufficiently to qualify as a partial response (PR) nor increased sufficiently to qualify as progressive disease (PD).
Complete Response Rate by RECIST v1.1 | 2 years
  Complete Response Rate assessed by RECIST v1.1. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) Complete Response (CR) is defined as the disappearance of all target lesions.
Partial Response Rate by RECIST v1.1 | 2 years
  Partial Response rate assessed by RECIST v1.1. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions

SECONDARY OUTCOMES:
Stable Disease Rate by RECIST v1.1 | 2 years
  Stable Disease Rate by RECIST v1.1. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD is defined as an increase of at least 20% in the sum of the longest diameters of the target lesions, with an absolute increase of at least 5 mm, or the appearance of one or more new lesions. Stable Disease (SD) is defined as a tumor that has neither shrunk sufficiently to qualify as a partial response (PR) nor increased sufficiently to qualify as progressive disease (PD).
Percentage of Responders by RECIST v1.1 | 2 years
  Sum of Complete Response (CR) + Partial Response (PR) to determine Percentage of Responders by RECIST v1.1. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions; Complete Response (CR) is defined as the disappearance of all target lesions. Percentage of Responders (POR) = CR + PR
Overall Survival | 2 years
  Survival rate of subjects who received at least one dose of Spedox-6.
Progression Free Survival | 2 years
  Survival rate of subjects who received at least one dose of Spedox-6 without Progression of their disease.
Number of Patients with Grade 3 non-hematological toxicities by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 2 years
  Number of Patients who received at least one dose of Spedox-6 with Grade 3 non-hematological toxicities (excluding alopecia) by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 version 5.0 with the following exceptions: Grade 3 nausea/vomiting or diarrhea <72 hours with adequate antiemetic and other supportive care; Grade 3 fatigue <1 week; Grade 3 electrolyte abnormality that lasts up to 72 hours, is not clinically complicated and resolves spontaneously or responds to conventional medical interventions.
Number of patients with Grade 4 non-hematologic (non-laboratory) by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 version 5.0 | 2 years
  Number of patients who received at least one dose of Spedox-6 with Grade 4 non-hematologic (non-laboratory) toxicity of any duration per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Number of patients with Grade 3 or Grade 4 febrile neutropenia by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 version 5.0 | 2 years
  Number of patients who received at least one dose of Spedox-6 with Grade 3 or Grade 4 febrile neutropenia of any duration per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Number of patients with Grade 3 Thrombocytopenia in Combination with Grade 3 or greater blood and lymphatic system disorder by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 version 5.0 | 2 years
  Number of patients who received at least one dose of Spedox-6 with Grade 3 Thrombocytopenia in Combination with Grade 3 or greater blood and lymphatic system disorder per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Number of patients with Grade 3 AST or ALT increase that is associated with a Grade 2 or greater Rise in Bilirubin by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 version 5.0 | 2 years
  Number of patients who received at least one dose of Spedox-6 with Grade 3 AST or ALT increase that is associated with a Grade 2 or greater Rise in Bilirubin per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

OTHER OUTCOMES:
Correlation between Tumor FcRn Expression (IHC Score) and Objective Response (per RECIST v1.1) | 2 years
  E valuate the correlation between tumor neonatal Fc receptor (FcRn) expression, as measured by immunohistochemistry (IHC) H-score, and objective tumor response, defined per RECIST v1.1 criteria (Complete Response or Partial Response).
Correlation between Tumor FcRn Expression (IHC Score) and Disease Control (CR + PR + SD per RECIST v1.1) | 2 years
  To evaluate the correlation between tumor neonatal Fc receptor (FcRn) expression, as assessed by immunohistochemistry (IHC) H-score, and disease control, defined as the proportion of patients achieving Complete Response (CR), Partial Response (PR), or Stable Disease (SD) per RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Chow, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No